CLINICAL TRIAL: NCT01886495
Title: High Protein Diet , Adiponectin and Inflammatory Factors
Brief Title: Effect of High Protein Diet on Adiponectin and Inflammation Among Overweight and Obese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Isfahan University of Medical Sciences, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: high protein diet in children
Record Dates: First submitted 2013-06-21; First posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Body Mass Index Quantitative Trait Locus 5 Disorder; Tangier Disease
MeSH Terms: conditions — Tangier Disease | interventions — Diet Therapy; Diet, High-Protein

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nutrition intervention (Active Comparator): high protein diet
  Interventions: Other: nutrition intervention
- control diet (No Intervention)

INTERVENTIONS:
Other: nutrition intervention
  Other Names: high protein diet
  Arms: nutrition intervention

SUMMARY:
The investigators aimed to determine the effects of HP diet on adiponectin and inflammatory factors among overweight and obese children.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 85th
* age of 6-11 years
* no history of chronic diseases
* taken medications

Exclusion Criteria:

* do not prescribe their diet
* mental retardation

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
adiponectin (mcg/ml) | 10 weeks
  amount of adiponectin

SECONDARY OUTCOMES:
interlukine 6 (mcg/ml) | 10 weeks
tumor necrosis factor alpha (ng/ml) | 10 weeks
C reactive protein (mcg/ml) | 10 weeks
fibrinogen (mcg/ml) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leila Azadbakht, PhD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Isfahan University of Medical Sciences Leila Azadbakht, Phd, Isfahan, Iran